CLINICAL TRIAL: NCT05866705
Title: The Mental Health Experiences of Sexual and Gender Minorities Living With Cancer and Their Care Partners
Acronym: SGMC
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Frank Puga, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300009168; PREP Award (Other: UAB Center for Palliative and Supportive Care)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Depression; Anxiety; Caregiver Burden; Stress; Chronic Illness
Keywords: cancer; mental health; LGBTQIA+
MeSH Terms: conditions — Depression; Anxiety Disorders; Caregiver Burden; Chronic Disease; Neoplasms; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer: Individuals living with cancer
- Care Partner: Care partner for someone who is living with cancer

SUMMARY:
The purpose of this study is to examine relationships between contextual stressors and stress moderators, depression symptom experience, resilience, frailty, and quality of life among older sexual gender minorities cancer survivors and their care partners.

DETAILED DESCRIPTION:
A priority focus in palliative care is supporting the well-being and mental health of older adults living with cancer and their care partners, particularly among populations carrying a disproportionate cancer burden, such as sexual and gender minorities (SGM). Previous reports indicate that SGMs experience increased cancer risk, less effective care, and poor outcomes than heterosexual, cis-gendered, and gender binary individuals. Thus, it is imperative to understand better the palliative and end-of-life (EOL) care needs of SGM cancer survivors and their care partners.

Recent studies have found that SGM individuals living with cancer report more depression than their heterosexual counterparts. These findings are concerning as increased distress and adverse mental health outcomes among individuals living with cancer have been shown to exacerbate symptom burden, impact disease progression, and increase the risk of suicide. Further, the care partners of SGM individuals living with cancer often serve as informal caregivers and may experience increased stress due to their loved one's diagnosis and disease progression. Such caregiving-related stress has been shown to increase the risk of late-life serious mental illness, accelerated aging, and age-related diseases. There is a critical need for culturally appropriate palliative care and EOL interventions that support the well-being of SGM individuals living with cancer and their care partners.

Further, limited knowledge exists on the relationship between daily and long-term patterns of psychological distress, specifically depression symptom experience, and changes in resilience (i.e., the capacity for positive adaptation despite adversity), frailty, and poor quality of life (QoL) over time. A failure to address this gap will result in continued health disparities in an underserved population in aging and palliative care.

ELIGIBILITY:
Inclusion Criteria

Individual living with cancer: 1) self-identifies as a sexual and/or gender minority; 2) ≥55 years of age; 3) diagnosed with cancer (stages 1 through 4), including brain, lung, breast, gynecologic, head and neck, gastrointestinal, genitourinary cancer, melanoma; and hematologic malignancies.

Care Partner: 1) ≥21 years of age; 2) self-identifies as a care partner of a sexual and/or gender minority diagnosed with cancer (stages 1 through 4), including brain, lung, breast, gynecologic, head and neck, gastrointestinal, genitourinary cancer, melanoma; and hematologic malignancies.

Exclusion Criteria

Individual living with cancer: 1) Medical documentation of active severe mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, suicidal ideation, uncorrected hearing loss, or substance abuse; 2) does not have reliable internet access.

Care Partner: 1) Self-reported mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse; 2) does not have reliable internet access.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: LGBTQIA+ Individuals living with cancer (aged 55+) and their care partners (aged 21+)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Daily Depression Symptom Experience | 28 days
  PROMIS Emotional Distress-Depression Short Form, a 4-item scale measuring common symptoms associated with depresison.
Daily Anxiety Symptom Experience | 28 days
  PROMIS Emotional Distress-Anxiety Short Form, a 4-item scale measuring common symptoms associated with anxiety.
Depression | 28 days
  PHQ-9, a 9-item scale for screening, diagnosing, monitoring and measuring the severity of depression.
Anxiety | 28 days
  GAD-7, a 7-item scale for screening, diagnosing, monitoring and measuring the severity of anxiety.

SECONDARY OUTCOMES:
Reslience | 28 days
  Resilience Scale for Adult: a 33-item scale measuring personal competence, social competence, personal structure, family coherence, and social support.
Health Related Quality of Life | 28 days
  PROMIS Global Health: 10 item scale measureing global health-related quality of life (HRQOL) across 2 domains: physical and mental health.
Fraility | 28 days
  Cancer & Aging Resilience Evaluation (CARE) Frailty Index: a 44-item scale that utilizes the principles of deficit accumulation to assess an individuals level of fraility.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Puga, Principal Investigator — University of Alabama at Birmingham School of Nursing
Locations (1):
- University of Alabama at Birmingham School of Nursing, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No